CLINICAL TRIAL: NCT04931914
Title: Antibiotic Regimens Tailored by Clinical Pharmacist Suppored by Intensivist Enhanced Rational Use of Antibiotics
Status: Completed | Type: Observational
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Ibrahim Mabrouk Ibrahim, lecturer in the anaesthesia department Alexandria university, University of Alexandria
Other Study IDs: 203
Record Dates: First submitted 2021-05-29; First posted 2021-06-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group c: Patients admitted from June 9, 2020 to june 31, 2021.
  Interventions: Other: Clinical pharmacy sharing in the patient care regimen

INTERVENTIONS:
Other: Clinical pharmacy sharing in the patient care regimen — antibiotic regimens will be directed by a trained clinical pharmacist recommendation and supported by intensivist.

SUMMARY:
adding pharmaceutical services to patient care and changing the professional activity of pharmacists from drug-focused to patient-oriented care,in the current study, clinical pharmacists will be assigned to monitor pharmacotherapy regimens, participate in patient care, and cooperate in educating the staff and evaluating care.

DETAILED DESCRIPTION:
During the intervention period, the pharmacist attended daily unit rounds with ICU intensivist with a focus on optimization of antibiotic regimens. Pharmacist consultative services were also available by phone calls 24 hours x 7 days if needed. For every patient surgical prophylactic antibiotic initiated immediately before surgery and continued for 48 hours following surgery. Antibiotic therapy had given as either directed or empiric. Directed therapy was defined as treatment of a documented infection based on culture and sensitivity. Empiric therapy was defined as any antibiotic therapy administered when no documented infection was present, and the patient had clinically suspected infection following surgery. Empiric antibiotic administration was required in majority of our SICU patients. Antibiotics had given after exclusion of allergy by history and intradermal sensitivity test.

ELIGIBILITY:
Inclusion Criteria:

* all admitted patients to the ICU between age 18-80 years old

Exclusion Criteria:

* Patient admitted for less than 24 hours (including deaths and transfers) will be excluded from the study.

Pediatric patients weighted less than kilograms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the information including the age, gender, comorbidity (presented as Charlson comorbidity index score ), surgical procedure done, patients' temperature, white blood cells count, type of infection (e.g., pneumonia, wound infection, Urinary tract infection,…..), prescribed antibiotics regimen either they will use empirical or based on cultures, results of culture sensitivity tests, length of stay, and mortality of patients
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Antibiotics consumption | 1 year
  consumption will be counted as number of defined daily doses (DDD), expressed as DDD per 100 patient-days
Average length of stay | 1 year
  the average number of days that patients spent in SICU.
Mortality rate | 1 year
  The number of deaths of patients admitted to SICU, divided by the number of admissions.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt